CLINICAL TRIAL: NCT00527800
Title: Interactions Between HIV and Malaria in African Children
Acronym: TCC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Makerere University (Other); The AIDS Support Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: CDC- PEPFAR CoAg#U62P024421
Record Dates: First submitted 2007-09-10; First posted 2007-09-11 (Estimated); Last update posted 2013-10-11 (Estimated); Status verified 2013-10

CONDITIONS: Malaria; HIV Infections
Keywords: Malaria; HIV; Trimethoprim-sulfamethoxazole; Artemether-lumefantrine; Dihydroartemisinin-piperaquine; Acute Infection
MeSH Terms: conditions — Malaria; HIV Infections | interventions — Artemether, Lumefantrine Drug Combination; Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Treatment for episodes of uncomplicated malaria
  Interventions: Drug: Dihydroartemisinin-piperaquine
- 2 (Active Comparator): Treatment for uncomplicated malaria
  Interventions: Drug: Artemether-lumefantrine
- A (Experimental): Prevention of malaria in HIV uninfected, exposed children
  Interventions: Drug: Trimethoprim-sulfamethoxazole
- B (No Intervention): Prevention of malaria in HIV uninfected, exposed children

INTERVENTIONS:
Drug: Dihydroartemisinin-piperaquine — Once daily for 3 days, given in fixed dose tablets (40 mg dihydroartemisinin + 320 mg piperaquine) according to weight-based guidelines
  Arms: 1
Drug: Artemether-lumefantrine — Dosed twice daily for 3 days, given in fixed dose tablets (20 mg artemether + 120 mg lumefantrine) according to weight-based guidelines
  Arms: 2
Drug: Trimethoprim-sulfamethoxazole — Once daily dosing according to weight based guidelines
  Arms: A

SUMMARY:
This is a prospective cohort study where HIV-infected and uninfected children will be enrolled between 6 weeks and 9 months of age and followed to the age of 21 months. All HIV-infected children will be given trimethoprim-sulfamethoxazole (TMP-SMX) prophylaxis as of 6 weeks of age. HIV-uninfected children born to HIV-infected mothers will be given TMP/SMX prophylaxis for the duration of breastfeeding and then randomized to the continuation of TMP/SMX or discontinuation of TMP/SMX prophylaxis. HIV-uninfected children born to HIV-uninfected mothers will not be given TMP/SMX prophylaxis. Study participants will be followed for all of their health care needs in a designated study clinic. All mother-child pairs will receive a basic care package including insecticide-treated bednets (ITNs) at enrollment. All HIV-infected mothers and children will receive antiretroviral therapy if eligible according to standardized World Health Organization (WHO) criteria. Study participants 4 months of age or older and at least 5 kg will be randomized to treatment with artemether-lumefantrine (AL) or dihydroartemisinin-piperaquine (DP) at the time of their first diagnosis of uncomplicated malaria. Study participants will receive the same antimalarial treatment regimen for all future episodes of uncomplicated malaria. Study participants less than 4 months of age or less than 5 kg diagnosed with malaria and all episodes of complicated malaria will be treated with quinine in accordance with local guidelines.

The investigators will test the hypotheses that:

1. TMP/SMX prophylaxis is highly effective in preventing malaria in both HIV-infected and HIV-uninfected children
2. The use of TMP/SMX prophylaxis is associated with an increased risk of infection with malaria parasites containing antifolate resistance-conferring mutations.
3. The use of antiretroviral (ARV) drugs is associated with a decreased incidence of malaria.
4. The efficacy, safety, and tolerability of AL and DP for the treatment of uncomplicated malaria differ.

   In 2008, we received approval and funding to extend the trial until 2012. We are now following all children through 5 years of age. First randomization to continue or discontinue TMP/SMX prophylaxis in our HIV-exposed population occurs 6-8 weeks after cessation of breastfeeding when HIV status can be confirmed as negative by DNA PCR. A second randomization occurs at 2 years of age in our HIV-exposed participants. At that point all HIV-exposed children who were originally randomized to continue TMP/SMX prophylaxis are again randomized to either immediately discontinue TMP/SMX prophylaxis or continue prophylaxis until age 4 years. All children will be off TMP/SMX between 4 and 5 years of age.

   We have also added an additional hypothesis to test during the study extension:
5. Prolonged TMP/SMX prophylaxis will result in an increased incidence of malaria in children in the year immediately following cessation of prophylaxis compared to children who have not used prophylaxis for over a year and those who have never been on prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

1. Age 6 weeks to 9 months
2. Documented HIV-1 status of mother and child
3. Agreement to come to the study clinic for any febrile episode or other illness
4. Agreement to avoid medications administered outside the study protocol
5. Guardian age 18 years or older (no age limit for parents)
6. Parent or guardian willing to provide informed consent
7. Residence within a 30 km radius of the study clinic

Exclusion Criteria:

1. HIV-exposed infants who have already stopped receiving TMP/SMX as a result of having stopped breastfeeding and having been tested HIV-negative before screening
2. Intention to move more than 30 km from the study clinic during the follow-up period
3. History of allergy or sensitivity to AL or DP or TMP/SMX
4. Active medical problem requiring in-patient evaluation at the time of screening

Ages: 6 Weeks to 9 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 351 (Actual)
Dates: Start 2007-08; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Incidence of clinical episodes of malaria | over entire course of follow-up
Risk of treatment failure at Day 28 defined as any early treatment failure or late clinical/parasitological failure adjusted and unadjusted by genotyping to distinguish recrudescence (treatment failure due to drug resistance) and new infections | 28 days following each malaria treatment

SECONDARY OUTCOMES:
Prevalence of mutations known to confer resistance to antifolate drugs in pretreatment samples from patients diagnosed with malaria | each time episode of malaria is diagnosed
Risk of adverse events | 28 days following each malaria treatment

CONTACTS AND LOCATIONS:
Overall Officials: Grant Dorsey, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Tororo District Hospital, Tororo, Uganda

REFERENCES:
- [Result] Creek DJ, Bigira V, McCormack S, Arinaitwe E, Wanzira H, Kakuru A, Tappero JW, Sandison TG, Lindegardh N, Nosten F, Aweeka FT, Parikh S. Pharmacokinetic predictors for recurrent malaria after dihydroartemisinin-piperaquine treatment of uncomplicated malaria in Ugandan infants. J Infect Dis. 2013 Jun 1;207(11):1646-54. doi: 10.1093/infdis/jit078. Epub 2013 Feb 27. PMID 23447696
- [Result] Kakuru A, Jagannathan P, Arinaitwe E, Wanzira H, Muhindo M, Bigira V, Osilo E, Homsy J, Kamya MR, Tappero JW, Dorsey G. The effects of ACT treatment and TS prophylaxis on Plasmodium falciparum gametocytemia in a cohort of young Ugandan children. Am J Trop Med Hyg. 2013 Apr;88(4):736-43. doi: 10.4269/ajtmh.12-0654. Epub 2013 Feb 4. PMID 23382157
- [Result] Jagannathan P, Muhindo MK, Kakuru A, Arinaitwe E, Greenhouse B, Tappero J, Rosenthal PJ, Kaharuza F, Kamya MR, Dorsey G. Increasing incidence of malaria in children despite insecticide-treated bed nets and prompt anti-malarial therapy in Tororo, Uganda. Malar J. 2012 Dec 28;11:435. doi: 10.1186/1475-2875-11-435. PMID 23273022
- [Result] Arinaitwe E, Gasasira A, Verret W, Homsy J, Wanzira H, Kakuru A, Sandison TG, Young S, Tappero JW, Kamya MR, Dorsey G. The association between malnutrition and the incidence of malaria among young HIV-infected and -uninfected Ugandan children: a prospective study. Malar J. 2012 Mar 27;11:90. doi: 10.1186/1475-2875-11-90. PMID 22453048
- [Result] Sandison TG, Homsy J, Arinaitwe E, Wanzira H, Kakuru A, Bigira V, Kalamya J, Vora N, Kublin J, Kamya MR, Dorsey G, Tappero JW. Protective efficacy of co-trimoxazole prophylaxis against malaria in HIV exposed children in rural Uganda: a randomised clinical trial. BMJ. 2011 Mar 31;342:d1617. doi: 10.1136/bmj.d1617. PMID 21454456
- [Result] Verret WJ, Arinaitwe E, Wanzira H, Bigira V, Kakuru A, Kamya M, Tappero JW, Sandison T, Dorsey G. Effect of nutritional status on response to treatment with artemisinin-based combination therapy in young Ugandan children with malaria. Antimicrob Agents Chemother. 2011 Jun;55(6):2629-35. doi: 10.1128/AAC.01727-10. Epub 2011 Mar 7. PMID 21383095
- [Result] Creek D, Bigira V, Arinaitwe E, Wanzira H, Kakuru A, Tappero J, Kamya MR, Dorsey G, Sandison TG. Increased risk of early vomiting among infants and young children treated with dihydroartemisinin-piperaquine compared with artemether-lumefantrine for uncomplicated malaria. Am J Trop Med Hyg. 2010 Oct;83(4):873-5. doi: 10.4269/ajtmh.2010.10-0158. PMID 20889882
- [Result] Vora N, Homsy J, Kakuru A, Arinaitwe E, Wanzira H, Sandison TG, Bigira V, Kamya MR, Tappero JW, Dorsey G. Breastfeeding and the risk of malaria in children born to HIV-infected and uninfected mothers in rural Uganda. J Acquir Immune Defic Syndr. 2010 Oct;55(2):253-61. doi: 10.1097/QAI.0b013e3181eb4fd7. PMID 20683193
- [Result] Katrak S, Gasasira A, Arinaitwe E, Kakuru A, Wanzira H, Bigira V, Sandison TG, Homsy J, Tappero JW, Kamya MR, Dorsey G. Safety and tolerability of artemether-lumefantrine versus dihydroartemisinin-piperaquine for malaria in young HIV-infected and uninfected children. Malar J. 2009 Nov 30;8:272. doi: 10.1186/1475-2875-8-272. PMID 19948038
- [Result] Arinaitwe E, Sandison TG, Wanzira H, Kakuru A, Homsy J, Kalamya J, Kamya MR, Vora N, Greenhouse B, Rosenthal PJ, Tappero J, Dorsey G. Artemether-lumefantrine versus dihydroartemisinin-piperaquine for falciparum malaria: a longitudinal, randomized trial in young Ugandan children. Clin Infect Dis. 2009 Dec 1;49(11):1629-37. doi: 10.1086/647946. PMID 19877969
- [Derived] Homsy J, Dorsey G, Arinaitwe E, Wanzira H, Kakuru A, Bigira V, Muhindo M, Kamya MR, Sandison TG, Tappero JW. Protective efficacy of prolonged co-trimoxazole prophylaxis in HIV-exposed children up to age 4 years for the prevention of malaria in Uganda: a randomised controlled open-label trial. Lancet Glob Health. 2014 Dec;2(12):e727-36. doi: 10.1016/S2214-109X(14)70329-8. PMID 25433628
- [Derived] Wanzira H, Kakuru A, Arinaitwe E, Bigira V, Muhindo MK, Conrad M, Rosenthal PJ, Kamya MR, Tappero JW, Dorsey G. Longitudinal outcomes in a cohort of Ugandan children randomized to artemether-lumefantrine versus dihydroartemisinin-piperaquine for the treatment of malaria. Clin Infect Dis. 2014 Aug 15;59(4):509-16. doi: 10.1093/cid/ciu353. Epub 2014 May 13. PMID 24825870
- [Derived] Conrad MD, LeClair N, Arinaitwe E, Wanzira H, Kakuru A, Bigira V, Muhindo M, Kamya MR, Tappero JW, Greenhouse B, Dorsey G, Rosenthal PJ. Comparative impacts over 5 years of artemisinin-based combination therapies on Plasmodium falciparum polymorphisms that modulate drug sensitivity in Ugandan children. J Infect Dis. 2014 Aug 1;210(3):344-53. doi: 10.1093/infdis/jiu141. Epub 2014 Mar 8. PMID 24610872
- [Derived] Muhindo MK, Kakuru A, Jagannathan P, Talisuna A, Osilo E, Orukan F, Arinaitwe E, Tappero JW, Kaharuza F, Kamya MR, Dorsey G. Early parasite clearance following artemisinin-based combination therapy among Ugandan children with uncomplicated Plasmodium falciparum malaria. Malar J. 2014 Jan 28;13:32. doi: 10.1186/1475-2875-13-32. PMID 24468007
- See also: MU-UCSF Research Collaboration website — http://www.muucsf.org/